CLINICAL TRIAL: NCT04837651
Title: A Real World, Prospective, Single-center, Observational Study Comparing Humoral and T-Cell Responses to COVID-19 Vaccination in Multiple Sclerosis Patients Treated With Ocrelizumab or Natalizumab
Brief Title: Humoral and T-Cell Responses to COVID-19 Vaccination in Multiple Sclerosis Patients Treated With Ocrelizumab Treated With Ocrelizumab or Natalizumab
Acronym: OCR-VAX
Status: Completed | Type: Observational
Sponsor: Dragonfly Research, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: VA26843
Record Dates: First submitted 2021-03-16; First posted 2021-04-08 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases; Autoimmune Diseases; Immune System Diseases; Pathologic Processes
Keywords: COVID-19; Natalizumab; Ocrelizumab; Ocrevus; Tysabri; Antibody; Coronavirus; Vaccine
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases; Autoimmune Diseases; Immune System Diseases; Pathologic Processes; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Ocrelizumab Treated Multiple Sclerosis Patients
  Interventions: Device: Elecsys semi-quantitative Anti-SARS-CoV-2 antibody test; Device: T-Detect COVID T-cell blood test
- Natalizumab Treated Multiple Sclerosis Patients
  Interventions: Device: Elecsys semi-quantitative Anti-SARS-CoV-2 antibody test; Device: T-Detect COVID T-cell blood test

INTERVENTIONS:
Device: Elecsys semi-quantitative Anti-SARS-CoV-2 antibody test — Subjects will receive an Elecsys semi-quantitative Anti-SARS-CoV-2 antibody test within 4 weeks of receiving their first COVID-19 injection. Within 3-4 weeks of receipt of their final COVID-19 vaccine dose, subjects will receive another Elecsys semi-quantitative Anti-SARS-CoV-2 antibody test.
Device: T-Detect COVID T-cell blood test — A select number of subjects will also receive a qualitative SARS-CoV-2 t-cell immunity test, the T-Detect COVID test, within 3-4 weeks of receipt of their final COVID-19 vaccine dose.

SUMMARY:
The primary goal of this study is to provide additional data regarding B and T-cell mediated responses to COVID-19 vaccines in MS patients treated with OCR and to determine which clinical and paraclinical variables correlating with vaccine immunogenicity. B-cell mediated humoral responses and adaptive T-cell mediated cellular responses were measured in patients treated with OCR who received any of the available SARS-CoV-2 vaccines, 3-4 weeks after completion of vaccination.

DETAILED DESCRIPTION:
The purpose of this study is to see if patients on ocrelizumab (Ocrevus) produce a humoral and T-cell response to the coronavirus vaccine. Ocrelizumab depletes B-lymphocytes and has the potential to reduce the effectiveness of vaccines. The impact of ocrelizumab treatment on coronavirus vaccines is unknown.

Natalizumab (Tysabri) likely has a minimal impact the efficacy of vaccines. In this study the investigators will take blood samples in patients being treated with either ocrelizumab or natalizumab before and after vaccination with an FDA-authorized coronavirus (COVID-19) vaccine and compare the antibody response in both groups.

ELIGIBILITY:
Inclusion Criteria

* Age 18-55
* Diagnosis of multiple sclerosis (as per the revised 2017 criteria)
* EDSS score of 0-5.5 inclusive
* Has initiated ocrelizumab or natalizumab at least 6 months prior to study enrollment
* For women of childbearing potential: agreement to remain abstinent or to use a highly effective (99% efficacy or greater) contraceptive method
* Individual must be able to provide consent, read/write/comprehend English language or must be able to provide a consistent translator

Exclusion Criteria

* Previous infection with COVID-19, confirmed by FDA approved testing
* Cognitive impairment limiting the ability to consent or complete study procedures
* Currently pregnant, planning to become pregnant during the study period, or currently breastfeeding
* Any prior use of immunosuppressive or chemotherapy treatment (including, but not limited to, cladribine, alemtuzumab, mycophenolate mofetil, cyclophosphamide, methotrexate, azathioprine)
* Prior treatment with a B-cell depleting therapy other than ocrelizumab within 12 months of first on-study infusion excluding standard ocrelizumab pre-treatment therapy
* Use of systemic corticosteroid therapy within 12 weeks of screening (excluding corticosteroid treatment given concurrently with ocrelizumab)
* History of allergic reactions to vaccines

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult Multiple Sclerosis patients receiving treatment with natalizumab or ocrelizumab at the Elliot Lewis MS Center.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 B-cell response | Measured within 3-4 weeks of final COVID-19 vaccine dose
  Production of SARS-CoV-2 antibodies in response to the COVID-19 vaccine in patients receiving treatment with ocrelizumab or natalizumab.
SARS-CoV-2 T-cell response | Measured within 3-4 weeks of final COVID-19 vaccine dose
  Production of SARS-CoV-2 T-cell response to the COVID-19 vaccine in patients receiving treatment with ocrelizumab or natalizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Katz, M.D., Principal Investigator — Dragonfly Research, LLC
Locations (1):
- Dragonfly Research, LLC, Wellesley, Massachusetts, United States